CLINICAL TRIAL: NCT01167855
Title: Reducing Asthma Disparities Through School-Based Telemedicine for Rural Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Arkansas Children's Hospital Research Institute (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); University of Arkansas (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 112695; 1R01HL102388-01 (NIH)
Record Dates: First submitted 2010-07-21; First posted 2010-07-22 (Estimated); Last update posted 2017-05-16 (Actual); Status verified 2017-05

CONDITIONS: Asthma; Quality of Life; Children
Keywords: Pediatric Asthma; Low-income; Arkansas Delta Region
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Intervention (Experimental): * Telemedicine asthma education sessions
  * Asthma health assessment via telemonitoring
  * Provider treatment prompts
  * School absenteeism
  * Prescription filling profile
  Interventions: Other: Asthma Education Sessions; Other: Asthma Health Assessment via Telemonitoring; Other: Provider Treatment Prompt; Other: School Absenteeism; Other: Prescription Filling Profile

INTERVENTIONS:
Other: Asthma Education Sessions — Comprehensive asthma education sessions delivered via telemedicine.
Other: Asthma Health Assessment via Telemonitoring — Each intervention participant will undergo assessment of asthma via school-based telemonitoring to measure lung function and provide a self-report of asthma symptoms.
Other: Provider Treatment Prompt — A treatment prompt will be mailed to the primary care provider at baseline and 3 months.
Other: School Absenteeism — Absenteeism before and after the intervention will be compared in the intervention group and also will be compared to absentee rates of the usual care group.
Other: Prescription Filling Profile — Study personnel will monitor participants' prescription profiles.

SUMMARY:
The overall goal of this proposal is to examine the efficacy of a school-based asthma telemedicine intervention in a predominately minority, low-income rural pediatric population.

DETAILED DESCRIPTION:
A total of 1110 subjects will be enrolled in this research study. Five hundred forty (540) subjects will be between the ages of 7-14 years. The remaining 540 subjects will be comprised of the primary caregiver of the participants. Thirty (30) school nurse/s providing care to the 270 intervention participants will also be enrolled in the study. To test our hypotheses, the investigators will conduct a cluster randomized trial with 540 children, ages 7-14 years and their parent/guardian(s), to address the following specific aims:

Specific Aim 1: Examine the efficacy of a school-based asthma telemedicine intervention in improving asthma-related health outcomes in an intervention group compared to children receiving usual care.

Specific Aim 2: Determine the effects of a school-based asthma telemedicine intervention on asthma self-management skills of intervention caregivers and participants compared to a usual care group. The investigators will compare changes in asthma self-efficacy, quality of life, and knowledge between groups.

Specific Aim 3: Determine the cost of the intervention in relation to health outcomes.

ELIGIBILITY:
Inclusion Criteria:

The investigators will recruit students (ages 7-14 years) with asthma who are currently enrolled in public school districts located in the Delta region of Arkansas.

Eligibility of identified children will be determined by a brief telephone survey. The survey questions will determine if the child fulfills inclusion/exclusion criteria.

1. Age ≥ 7 and ≤ 14 years.
2. Use of asthma medications for acute relief of symptoms (rescue) or for control of symptoms (preventive) in the past 6 months. Children not on a controller who report using a rescue medication only for prevention of exercised-induced symptoms will not be eligible for the study.
3. Physician-diagnosed asthma by parent/caregiver report. OR
4. In the absence of a formal physician diagnosis, the caregiver must report symptoms consistent with at least mild persistent asthma. The investigators will use asthma screening criteria to ensure that participants meet eligibility requirements. Participants must establish a history of episodic airflow obstruction or airway hyperresponsiveness and meet National Heart Lung and Blood Institute (NHLBI) guidelines for persistent asthma. Mild persistent asthma will be defined as any 1 of the following during the prior 4 weeks (by caregiver report):

   * An average of > 2 days per week with asthma symptoms
   * > 2 days per week with rescue medication use
   * > 2 nights per month awakened with nighttime symptoms
   * Minor limitation of activity
   * ≥ 2 episodes of asthma during the past year that have required systemic corticosteroids

Exclusion Criteria:

1. Significant underlying respiratory disease other than asthma (such as cystic fibrosis or chronic lung disease) that could potentially interfere with asthma-related outcome measures.
2. Significant co-morbid conditions (such as severe developmental delay) that could preclude participation in an education-based intervention.
3. Inability to speak or understand English (child or parent).
4. Children in foster care or other situations in which consent cannot be obtained from a guardian.
5. Prior enrollment in the study.
6. Families without access to a working telephone as all survey data will be collected via telephone.

Ages: 7 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 823 (Actual)
Dates: Start 2011-05-25 (Actual); Primary Completion 2017-02-01 (Actual); Study Completion 2017-02-01 (Actual)

PRIMARY OUTCOMES:
Symptom Free Days | The number of symptom-free days (SFD) during the prior 2 weeks assessed at the end of the intervention.
  Examine the efficacy of a school-based asthma telemedicine intervention.

SECONDARY OUTCOMES:
Secondary Clinical Outcomes | Secondary outcomes will be measured during the intervention, at the end of the intervention and at 6-month follow-up.
  Secondary clinical outcomes will be measured at specific time points during the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Tamara T. Perry, M.D., Principal Investigator — University of Arkansas
Locations (1):
- Arkansas Children's Hospital Research Institute, Little Rock, Arkansas, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to share individual participant data.

REFERENCES:
- [Background] Perry TT, Vargas PA, McCracken A, Jones SM. Underdiagnosed and uncontrolled asthma: findings in rural schoolchildren from the Delta region of Arkansas. Ann Allergy Asthma Immunol. 2008 Oct;101(4):375-81. doi: 10.1016/S1081-1206(10)60313-4. PMID 18939725
- [Background] Pesek R, PA V, Jones S, McCracken A, Perry TT. Pediatric asthma diagnosis and morbidity in urban and rural Arkansas. J Allergy Clin Immunol 2009;123:S210.
- [Background] Vargas PA, Simpson PM, Gary Wheeler J, Goel R, Feild CR, Tilford JM, Jones SM. Characteristics of children with asthma who are enrolled in a Head Start program. J Allergy Clin Immunol. 2004 Sep;114(3):499-504. doi: 10.1016/j.jaci.2004.05.025. PMID 15356547
- [Background] Tilford JM. Cost-effectiveness analysis and emergency medical services for children: issues and applications. Ambul Pediatr. 2002 Jul-Aug;2(4 Suppl):330-6. doi: 10.1367/1539-4409(2002)0022.0.co;2. PMID 12135408
- [Derived] Perry TT, Halterman JS, Brown RH, Luo C, Randle SM, Hunter CR, Rettiganti M. Results of an asthma education program delivered via telemedicine in rural schools. Ann Allergy Asthma Immunol. 2018 Apr;120(4):401-408. doi: 10.1016/j.anai.2018.02.013. Epub 2018 Feb 19. PMID 29471032